CLINICAL TRIAL: NCT01862120
Title: Induction of Regulatory T Cells for the Treatment of Recently Diagnosed Type 1 Diabetes: Dose Finding Study of the Lowest Active Dose of IL-2 in Children
Brief Title: Dose Finding Study of Il-2 at Ultra-low Dose in Children With Recently Diagnosed Type 1 Diabetes
Acronym: DFIL2-Child
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P101106
Record Dates: First submitted 2012-12-10; First posted 2013-05-24 (Estimated); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Type 1 Diabetes
Keywords: Recently diagnosed; Regulatory T Cells; Tolerance Induction; Paediatrics; Low dose; IL-2
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- interleukin-2 (Experimental): Dose D1 of interleukin-2
  Interventions: Drug: Dose D1 of interleukin-2
- Dose D2 of interleukin-2 (Experimental): Dose D2 of interleukin-2
  Interventions: Drug: Dose D2 of Interleukin-2
- Dose D3 of interleukin-2 (Experimental): Dose D3 of interleukin-2
  Interventions: Drug: Dose D3 of interleukin-2
- placebo (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Dose D1 of interleukin-2 — subcutaneous injection of Interleukin-2 during 5 days, once daily repeated administration(Induction period). At day 15 single administration of Interleukin-2 every two weeks during one year (maintenance period).
  Arms: interleukin-2
Drug: placebo — subcutaneous injection of Interleukin-2 during 5 days, once daily repeated administration(Induction period). At day 15 single administration of Interleukin-2 every two weeks during one year (maintenance period).
  Arms: placebo
Drug: Dose D2 of Interleukin-2 — subcutaneous injection of Interleukin-2 during 5 days, once daily repeated administration(Induction period). At day 15 single administration of Interleukin-2 every two weeks during one year (maintenance period).
  Arms: Dose D2 of interleukin-2
Drug: Dose D3 of interleukin-2 — subcutaneous injection of Interleukin-2 during 5 days, once daily repeated administration(Induction period). At day 15 single administration of Interleukin-2 every two weeks during one year (maintenance period).
  Arms: Dose D3 of interleukin-2

SUMMARY:
Human recombinant interleukin-2 (rhIL-2) is a biological signalling protein playing a key role in the regulation of the immune system. At high doses, rhIL-2 activates the immune effectors T cells (TEFFS) while at low doses rhIL-2 induces and activates regulatory T cells (TREGS), a population of immune cells controlling the immune Teff response. In patients with Type 1 Diabetes (T1D), TREGS fail to control the autoimmune destruction by TEFFS of pancreatic beta-cells producing insulin. The investigator recently showed that rhIL-2 at low dose is well tolerated in patients with an autoimmune disease and in adults with established T1D, inducing TREGS without effects on TEFFS. The investigators aim to use rhIL-2 at low dose to induce/stimulate TREGS in young recently diagnosed T1D patients. This study will investigate the dose effect relationship of low dose rhIL-2 on TREG induction such as to optimize the risk benefit ratio of this treatment in T1D. Through Treg induction, the investigators aim to protect the remaining/regenerating pancreatic β-cells from autoimmune destruction, thus improving or even curing T1D.

DETAILED DESCRIPTION:
Main objective:

Define the lowest dose of rhIL-2 inducing TREGS in children with recently diagnosed type 1 diabetes.

Conduct of the study:

Three doses will be studied versus placebo in parallel groups of six patients. Each dose or placebo will be studied according to three periods of treatment:

1. Induction of TREGS following a cure of 5 days repeated once daily administration [day 1 - day 5].
2. Maintenance of TREGS following repeated administration once every two weeks for one year [day 15 - day 337].

At each treatment period, Treg response and tolerance will be evaluated. In addition, overall response on T1D parameters will be assessed throughout the study.

ELIGIBILITY:
Inclusion criteria :

* Age [7-13] years for girls and [7-14] years for boys

  * With a T1D diagnosis (as ADA)
  * Treated with insulin for ≤ 3 months,
  * With at least one auto-antibody among: anti-insulin, anti-GAD, anti-IA2, anti-ZnT8 ;
* No clinically relevant abnormal findings for haematology, biochemistry, liver and kidney functions
* Informed consent signed by the patient, the parents, and the investigator before any intervention necessary for the trial.

Exclusion criteria :

* Contra-indications to IL-2 :

  * Hyper sensibility to IL-2 or its excipients,
  * Severe cardiopathy
  * Previous organ allograft
  * Ongoing infection requiring antibiotherapy,
  * O2 Saturation ≤ 90 %
  * Severe impairment of any vital organ
  * Documented history of other auto-immune diseases (except for auto-antibodies for, IAA, GADA, IA-2A, anti-ZnT8A, and stable thyroiditis with normal TSH (<10 mUI/L), T3 and, T4 levels.
  * Diabetes onset characteristics including:

    * Continuous nocturnal polyuria ≥ 3 months ;
    * Inaugural acidosis (with venous Ph < 7.25) ;
    * HbA1c at diagnostic ≥ 13%;
    * Weight loss ≥ 10 % at diagnosis ;
    * Positive autoantibodies to 21-hydroxylase
    * Stage 2 obesity
* Non authorized concomitant treatment : immuno-modulators, cytotoxic drugs, drug modifying plasma glycemia
* vaccination ≤ 4 weeks with life vaccin
* Positive serology (IgM) to the Epstein-Barr virus (EBV) and/or cytomegalovirus (CMV), reflecting an acute infection.
* Participation to another clinical investigation in previous 3 months
* No affiliation to National Health Insurance

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2013-06-27 (Actual); Primary Completion 2016-07-08 (Actual); Study Completion 2017-03-16 (Actual)

PRIMARY OUTCOMES:
Treg response following the induction cure period | day 5
  expressed as % total CD4 cells

SECONDARY OUTCOMES:
Fasting plasma concentration of C-peptide | at Day 0, 99, 183, 267, 351, 436
C-peptide AUC response to a mixed meal tolerance test | at baseline, at months 6, 12, 15
IDAA1C score | at baseline, at months 3, 6, 9, 12, 15
  is a score defined as A1C (percent) + [4 x insulin dose (units per kilogram per 24 h)] without unit
HbA1c | at baseline, at months 3, 6, 9, 12, 15
Treg response after the last administration | day 351, day 436
Treg response during the maintenance period compare to the baseline | day 15, day 29, day 43, day 99, day 183, day 267
  Treg response expressed as the % / CD4 will be measured several times

CONTACTS AND LOCATIONS:
Overall Officials: David Klatzmann, MD, PhD, Principal Investigator — APHP
Locations (6):
- France (6):
  - Service d'Endocrinologie Pédiatrique, Le Kremlin-Bicêtre
  - Service de Pédiatrie - CHU de Nîmes, Nîmes
  - CIC pédiatrique - CHU de Necker, Paris
  - Service d'endocrinologie pédiatrique - CHU de Necker, Paris
  - CIC 9202 CHU Rober Débré, Paris
  - Service d'endocrinologie Diabétologie pédiatrique CHU Robert Débré, Paris

REFERENCES:
- [Derived] Rosenzwajg M, Salet R, Lorenzon R, Tchitchek N, Roux A, Bernard C, Carel JC, Storey C, Polak M, Beltrand J, Amouyal C, Hartemann A, Corbeau P, Vicaut E, Bibal C, Bougneres P, Tran TA, Klatzmann D. Low-dose IL-2 in children with recently diagnosed type 1 diabetes: a Phase I/II randomised, double-blind, placebo-controlled, dose-finding study. Diabetologia. 2020 Sep;63(9):1808-1821. doi: 10.1007/s00125-020-05200-w. Epub 2020 Jul 1. PMID 32607749